CLINICAL TRIAL: NCT02451267
Title: Clinical Prediction Rule for Identifying Patients With Chronic Neck Pain Who Will Benefit From General Aerobic Exercise
Brief Title: Clinical Prediction Rules for Identifying Patients With Chronic Neck Pain Who Will Benefit From General Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, Prof. Refael Carel, Professor, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COM-0016-15
Record Dates: First submitted 2015-05-10; First posted 2015-05-21 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Neck Pain
Keywords: neck pain; aerobic exercise; cervical pain
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- positive CPR: research group (Experimental): physical therapy treatment with aerobic exercise
  Interventions: Other: physical therapy treatment with aerobic exercise
- negative CPR: research group (Experimental): physical therapy treatment with aerobic exercise
  Interventions: Other: physical therapy treatment with aerobic exercise
- positive CPR: control group (Active Comparator): physical therapy treatment
  Interventions: Other: physical therapy treatment
- negative CPR: control group (Active Comparator): physical therapy treatment
  Interventions: Other: physical therapy treatment

INTERVENTIONS:
Other: physical therapy treatment with aerobic exercise — neck exercise strengthening program with neck massage and aerobic exercise (leg bicycling with relaxed shoulders)
  Arms: negative CPR: research group; positive CPR: research group
Other: physical therapy treatment — neck exercise strengthening program with neck massage
  Arms: negative CPR: control group; positive CPR: control group

SUMMARY:
The aim of the study is to investigate the effect of aerobic exercise on chronic neck pain. The study will be double blind randomized controlled trial . 120 patients with neck pain will be recruited for the study and divided into a research group and control group. The research group will receive neck exercise program with neck massage and aerobic exercise (leg bicycling with relaxed shoulders) and the control group will receive only neck exercise program with neck massage. Both intervention will be delivered by physiotherapist over 10 treatments and will include a home exercise program. In addition, clinical prediction rule (CPR) for identifying patients with neck pain who will respond better to an aerobic treatment program will be defined.

DETAILED DESCRIPTION:
Background:Recently, Hanney et al (2013) derived a preliminary clinical prediction rule (CPR) for identifying patients with neck pain (NP) who may respond to an exercise-based treatment program. These CPRs of neck exercise has not considered aerobic exercise (AE) on NP treatment.

Aims of this study: 1) To investigate the effect of aerobic exercise on chronic neck pain;2) To derive a clinical prediction rule for identifying patients with neck pain who may benefit from aerobic treatment program; 3) To determine the prevalence of neck pain in Israel.

Study Design: Double Blind Randomized controlled trial setting: Outpatients physical therapy clinics of "Clalit Health Services" in Haifa and Western Galilee area.

Participants: Patients referred to physical therapy with a primary diagnosis of chronic non-specific NP.

Methods: Following a baseline examination in which the subjects' status on the CPR will be determined, the subjects (CPR positive and negative) will be randomized, divided into a research group and control group. The CPR status will be determined according to Hanney's paper (e.g.: neck disability Index score < 18/50 ,shoulder protraction, cervical side bending < 32°,Fear avoidance belief questionnaire-physical activity score < 15, not active on a regular basis on bicycle training). Positive CPR is accordance of having 4/5 these points.

The baseline examination will include: active and passive cervical range of motion, neurological exam (reflex, sensation, muscle testing), cervical segmental mobility (accessory movement), neck muscle length, cervical manual muscle test and posture assessment.

The research group will receive neck exercise program with neck massage and AE (leg bicycling with relaxed shoulders) and the control group will receive neck exercise program with neck massage. Both intervention will be delivered by physiotherapist over 10 treatments and will include a home exercise program. Immediate examination will be used at the last treatment (10 treatments), and at 3 and 6 month follow up examination for long-term effects.

In addition, Data collecting from physiotherapy department in "Clalit Health Services" about statistic of patients with NP who referred to physical therapy including: Prevalence, demographic and profile data

ELIGIBILITY:
Inclusion Criteria:

* chronic neck pain (> 30 days)
* neck disability index >10
* not physical active on a daily basis

Exclusion Criteria:

* past history of whiplash injury or cervical surgery
* pain radiates to the upper limb with neurological deficit (reduced reflex, sensation, muscle strength)
* complain of vertigo
* cervical spine diseases: Spondylosis, Spondylolisthesis

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Global Rating of Change (GROC) scale | following 6 weeks of treatment, 3 months and 6 months
  rating pain severity on a scale from -7 to 7

SECONDARY OUTCOMES:
Change from baseline in Neck Disability Index at 6 weeks | following 6 weeks of treatment
  Questionnaire assessing the individuals disability due to the neck pain
Change from baseline in Fear Avoidance Beliefs Questionnaire | following 6 weeks of treatment
  Questionnaire about the individuals fear that his pain is caused due to movement or work
Change from baseline in cervical range of motion | following 6 weeks of treatment
  active range of motion using inclinometer
long term follow up assessment of VAS | 3 months and 6 months
  phone assessment of cervical pain severity
long term follow up assessment Neck Disability Index | 3 months and 6 months
  phone assessment of individuals disability
Change from baseline in Visual Analog Scale (VAS) at 6 weeks | following 6 weeks of treatment
  rating pain severity on a scale from 0-10
headache complaints | following 6 weeks of treatment, 3 months and 6 months
  complains of headache episodes
medication consumption for pain relief | following 6 weeks of treatment, 3 months and 6 months
  how many medication the patient used

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Study Director — University of Haifa, Department of Physical Therapy
Locations (1):
- Clalit Health Service, Nazareth, Israel

REFERENCES:
- [Background] Hanney WJ, Kolber MJ, George SZ, Young I, Patel CK, Cleland JA. Development of a preliminary clinical prediction rule to identify patients with neck pain that may benefit from a standardized program of stretching and muscle performance exercise: a prospective cohort study. Int J Sports Phys Ther. 2013 Dec;8(6):756-76. PMID 24377062
- [Background] Holth HS, Werpen HK, Zwart JA, Hagen K. Physical inactivity is associated with chronic musculoskeletal complaints 11 years later: results from the Nord-Trondelag Health Study. BMC Musculoskelet Disord. 2008 Dec 1;9:159. doi: 10.1186/1471-2474-9-159. PMID 19046448
- [Derived] Daher A, Dar G, Carel R. Effectiveness of combined aerobic exercise and neck-specific exercise compared to neck-specific exercise alone on work ability in neck pain patients: a secondary analysis of data from a randomized controlled trial. Int Arch Occup Environ Health. 2021 Oct;94(7):1739-1750. doi: 10.1007/s00420-021-01684-0. Epub 2021 Mar 17. PMID 33730206